CLINICAL TRIAL: NCT00621504
Title: A Phase 3, Multicenter, Randomized, Double-blind, Comparative Study to Evaluate the Safety and Efficacy of Ceftaroline Versus Ceftriaxone, With Adjunctive Clarithromycin, in the Treatment of Adult Subjects With Community-Acquired Pneumonia
Brief Title: Comparative Study of Ceftaroline vs. Ceftriaxone in Adult Subjects With Community-Acquired Pneumonia
Acronym: CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P903-08
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Pneumonia
Keywords: ceftaroline; Community-acquired pneumonia; CAP; IV (intravenous); Streptococcus pneumoniae; Haemophilus influenzae; Mycoplasma pneumoniae; Chlamydophila spp; Legionella spp; Multi-drug resistant Streptococcus pneumoniae (MDRSP); antimicrobial resistance; pneumococci; Ceftriaxone; bacteria; ß-lactam; beta-lactam; antibiotic
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Pneumonia; Haemophilus Infections | interventions — Ceftaroline; Injections; Ceftriaxone; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline fosamil for Injection (Experimental): Ceftaroline fosamil was administered in two consecutive 300-mg IV infusions over 30 minutes, every 12 hours (q12h).
  In both treatment groups, two doses of oral clarithromycin (500 mg q12h), defined as adjunctive therapy, were initiated on Study Day 1 with study drug therapy in order to provide an immunomodulatory benefit and initial therapy for possible infection due to an atypical organism.
  Interventions: Drug: Ceftaroline fosamil for Injection; Drug: Clarithromycin
- IV Ceftriaxone (Active Comparator): Ceftriaxone was administered as a 1-g IV infusion over 30 minutes followed by IV saline placebo infused over 30 minutes, every 24 hours (q24h).
  In both treatment groups, two doses of oral clarithromycin (500 mg q12h), defined as adjunctive therapy, were initiated on Study Day 1 with study drug therapy in order to provide an immunomodulatory benefit and initial therapy for possible infection due to an atypical organism.
  Interventions: Drug: IV Ceftriaxone; Drug: Placebo; Drug: Clarithromycin

INTERVENTIONS:
Drug: Ceftaroline fosamil for Injection — 2 consecutive, 300 mg dose parenteral infused over 30 minutes, every 12 hours, for 5 to 7 days
  Arms: Ceftaroline fosamil for Injection
Drug: IV Ceftriaxone — 1 g dose parenteral infused over 30 minutes, every 24 hours, for 5 to 7 days
  Other Names: Ceftriaxone
  Arms: IV Ceftriaxone
Drug: Placebo — Subjects randomized to receive ceftriaxone will receive ceftriaxone at a dose of 1 g infused over 30 minutes followed by IV saline placebo infused over 30 minutes, every 24 hours (q24h). Twelve hours after each dose of ceftriaxone and saline placebo (ie, between ceftriaxone doses), subjects in this group will receive two consecutive saline placebo infusions, each infused over 30 minutes q24h. The ceftriaxone and saline placebo infusions will correspond to the q12h infusions of ceftaroline, thereby maintaining the blind
  Arms: IV Ceftriaxone
Drug: Clarithromycin — In both treatment groups, two doses of oral clarithromycin (500 mg q12h), defined as adjunctive therapy, were initiated on Study Day 1 with study drug therapy in order to provide an immunomodulatory benefit and initial therapy for possible infection due to an atypical organism.

SUMMARY:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of Community-Acquired Pneumonia

DETAILED DESCRIPTION:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of Community-Acquired Pneumonia. Clinical trials for this study is held in many countries

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet the following inclusion criteria:

* Community-acquired pneumonia
* initial hospitalization, or treatment in an emergency room or urgent care setting
* infection would require initial treatment with IV antimicrobials.

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

* CAP suitable for outpatient therapy with an oral antimicrobial agent
* respiratory tract infections not due to community-acquired bacterial
* Non-infectious causes of pulmonary infiltrates
* Pleural empyema
* Infection with an atypical organism
* History of any hypersensitivity or allergic reaction to any ß-lactam antimicrobial
* History of any hypersensitivity or allergic reaction to clarithromycin or any macrolide/ ketolide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M File, MD, MS, Study Director — Summa Health System
Locations (133):
- United States (12):
  - Investigational site, Los Angeles, California
  - Investigational Site, Pasadena, California
  - Investigational Site, Sacramento, California
  - Investigational Site, San Diego, California
  - Investigational Site, Orlando, Florida
  - Investigational Site, Fort Gordon, Georgia
  - Investigational Site, Peoria, Illinois
  - Investigational Site, Baltimore, Maryland
  - Investigational site, Minneapolis, Minnesota
  - Investigational Site, Butte, Montana
  - Investigational Site, Akron, Ohio
  - Investigational Site, Houston, Texas
- Argentina (4):
  - Investigational Site, Buenos Aires, C.a.b.a.
  - Investigational Site, San Miguel de Tucumán, Tucumán Province
  - Investigational Site, Buenos Aires
  - Investigational Site, Vicente López
- Investigational Site, Vienna, Austria
- Brazil (10):
  - Investigational Site, Goiânia, G.o.
  - Investigational Site, Porto Alegre, Rio Grande do Sul
  - Investigational Site, São José do Rio Preto, São Paulo
  - Investigational Site 2, Belo Horizonte
  - Investigational Site 1, Belo Horizonte MG
  - Investigational Site, Campinas
  - Investigational Site, Curitiba-PR
  - Investigational Site, Juiz de Fora
  - Investigational site, Porto Alegre
  - Investigational Site, São Paulo
- Bulgaria (3):
  - Investigational Site, Burgas
  - Investigational Site, Sofia
  - Investigational Site, Varna
- Estonia (2):
  - Investigational Site, Tallinn
  - Investigational Site, Tartu
- France (3):
  - Investigational Site, Annecy
  - Investigational Site, Argenteuil
  - Investigational Site, Paris
- Investigational Site, Tbilisi, Georgia
- Germany (12):
  - Investigational Site, Lindenberger, State of Berlin
  - Investigational Site, Berlin
  - Investigational Site, Bochum
  - Investigational Site, Erfurt
  - Investigational Site, Heppenheim an der Bergstrasse
  - Investigational Site, Lich
  - Investigational Site, Lübeck
  - Investigational Site, Lüdenscheid
  - Investigational Site, Paderborn
  - Investigational Site, Schkeuditz
  - Investigational Site, Ulm
  - Investigational Site, Wiesbaden
- Hungary (8):
  - Investigational Site, Tatabánya, Szanatorium
  - Investigational Site, Budapest
  - Investigational Site, Mátraháza
  - Investigational Site, Miskolc
  - Investigational Site, Pécs
  - Investigational Site, Sopron
  - Investigational Site, Tatabánya
  - Investigational Site, Törökbálint
- Investigational Site, Vellore, Tamil Nadu, India
- Lithuania (4):
  - Investigational Site, Kaunas
  - Investigational Site, Klaipėda
  - Investigational Site, Šiauliai
  - Investigational Site, Vilnius
- Malaysia (5):
  - Investigational Site, Johor Bahru, Johor
  - Inestigational Site, Cheras, Kuala Lumpur
  - Investigational Site, George Town, Pulau Pinang
  - Investigational Site, Kedah
  - Investigational Site, Kuala Lumpur
- Poland (12):
  - Investigational Site, Będzin
  - Investigational Site, Brzesku
  - Investigational Site, Bytom
  - Investigational Site, Chodzież
  - Investigational Site, Częstochowa
  - Investigational Site, Katowice-Ochojec
  - Investigational Site, Krakow
  - Investigational Site, Lublin
  - Investigational Site, Poznan
  - Investigational Site, Tychy
  - Investigational Site, Warsaw
  - Investigational Site, Wroclaw
- Romania (8):
  - Inestigational Site, Bucharest
  - Investigational Site, Bucharest
  - Investigational Site, Cluj-Napoca
  - Investigational Site, Constanța
  - Investigational Site, Oradea
  - Investigational Site, Saint Brasov
  - Investigational Site, Târgu Mureş
  - Investigational Site, Timișoara
- Russia (8):
  - Investigational Site, Petrozavodsk, Republic of Karelia
  - Investigational Site, Arkhangelsk
  - Investigational Site, Moscow
  - Investigational Site, Rostov-on-Don
  - Investigational Site, Saint Petersburg
  - Investigational Site, Saratov
  - Investigational Site, Tatarstan
  - Investigational Site, Yekaterinburg
- Serbia (3):
  - Investigational Site, Belgrade
  - Investigational Site, Knez-Selo
  - Investigational Site, Kragujevac
- Slovakia (2):
  - Investigational Site, Bratislava
  - Slovakia, Nitra-Zobor
- South Africa (8):
  - Investigational Site, Bellville, Capetown
  - Investigational Site, Benomi
  - Investigational Site, Cape Town
  - Investigational Site, Krugersdorp
  - Investigational Site, Port Elizabeth
  - Investigational Site, Pretoria
  - Investigational Site, Somerset West
  - Investigational Site, Worcester
- Spain (6):
  - Investigational Site, Barcelona
  - Investigational Site, Elche
  - Investigational Site, León
  - Investigational Site, Madrid
  - Investigational Site, Valencia
  - Investigational Site, Vizcaya
- Switzerland (4):
  - Investigational Site, Biel
  - Investigational Site, Geneva
  - Investigational Site, La Chaux-de-Fonds
  - Investigational Site, Lugano
- Thailand (5):
  - Investigational Site, Bangkok
  - InvestigationalSite, Bangkok
  - Investigational Site, Chiang Mai
  - Investigational Site, Khonkaen
  - Investigational Site, Nonthaburi
- Ukraine (11):
  - Investigational Site, Aviv
  - Investigational Site, Dnipropetrovsk
  - Investigational Site, Donetsk
  - Investigational Site, Ivano-Frankivsk
  - Investigational Site, Kharkiv
  - Inestigational Site, Kyiv
  - Investigational Site, Kyiv
  - Investigational Site, Luhansk
  - Investigational Site, Odesa
  - Investigational Site, Poltava
  - Investigational Site, Uzhhorod

REFERENCES:
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Taboada M, Melnick D, Iaconis JP, Sun F, Zhong NS, File TM, Llorens L, Friedland HD, Wilson D. Ceftaroline fosamil versus ceftriaxone for the treatment of community-acquired pneumonia: individual patient data meta-analysis of randomized controlled trials. J Antimicrob Chemother. 2016 Apr;71(4):862-70. doi: 10.1093/jac/dkv415. Epub 2015 Dec 24. PMID 26702925
- [Derived] Lodise TP, Anzueto AR, Weber DJ, Shorr AF, Yang M, Smith A, Zhao Q, Huang X, File TM. Assessment of time to clinical response, a proxy for discharge readiness, among hospitalized patients with community-acquired pneumonia who received either ceftaroline fosamil or ceftriaxone in two phase III FOCUS trials. Antimicrob Agents Chemother. 2015 Feb;59(2):1119-26. doi: 10.1128/AAC.03643-14. Epub 2014 Dec 8. PMID 25487791
- [Derived] Shorr AF, Kollef M, Eckburg PB, Llorens L, Friedland HD. Assessment of ceftaroline fosamil in the treatment of community-acquired bacterial pneumonia due to Streptococcus pneumoniae: insights from two randomized trials. Diagn Microbiol Infect Dis. 2013 Mar;75(3):298-303. doi: 10.1016/j.diagmicrobio.2012.12.002. Epub 2013 Jan 26. PMID 23357290
- [Derived] Rank DR, Friedland HD, Laudano JB. Integrated safety summary of FOCUS 1 and FOCUS 2 trials: Phase III randomized, double-blind studies evaluating ceftaroline fosamil for the treatment of patients with community-acquired pneumonia. J Antimicrob Chemother. 2011 Apr;66 Suppl 3:iii53-9. doi: 10.1093/jac/dkr099. PMID 21482570
- [Derived] File TM Jr, Low DE, Eckburg PB, Talbot GH, Friedland HD, Lee J, Llorens L, Critchley IA, Thye DA; FOCUS 1 investigators. FOCUS 1: a randomized, double-blinded, multicentre, Phase III trial of the efficacy and safety of ceftaroline fosamil versus ceftriaxone in community-acquired pneumonia. J Antimicrob Chemother. 2011 Apr;66 Suppl 3:iii19-32. doi: 10.1093/jac/dkr096. PMID 21482566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was from 02 January 2008 to 29 December 2008
Pre-assignment Details: Patients were screened for up to 24 hours
Groups:
- Ceftaroline Fosamil for Injection: Ceftaroline fosamil was administered in two consecutive 300-mg IV infusions over 30 minutes, every 12 hours (q12h)
- IV Ceftriaxone: Ceftriaxone was administered as a 1-g IV infusion over 30 minutes followed by IV saline placebo infused over 30 minutes, every 24 hours (q24h).
Period: Overall Study
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Started | 299 | 307
Completed | 273 | 282
Not Completed | 26 | 25
Not completed — Adverse Event | 1 | 3
Not completed — At the request of sponsor/investigator | 1 | 0
Not completed — Withdrew consent | 9 | 6
Not completed — Lost to Follow-up | 8 | 10
Not completed — Other | 1 | 0
Not completed — Death | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone | Total
Number analyzed (Participants) | 299 | 307 | 606
Age, Customized [Number; unit: participants]
  <65 years | 154 | 157 | 311
  >= 65 years | 145 | 150 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (16.6) | 61.0 (16.6) | 61.0 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 112 | 220
  Male | 191 | 195 | 386
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 29 | 27 | 56
  Non-Hispanic | 270 | 280 | 550

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate at Test-of-Cure (TOC) in the Modified Intent-to-Treat Efficacy (MITTE) Populations
Description: Cure:Total resolution of all signs and symptoms of pneumonia (ie,CABP), or improvement to such an extent that further antimicrobial therapy was not necessary
  Failure: Any of the following:
  * Persistence, incomplete clinical resolution, or worsening in signs and symptoms of CABP that required alternative antimicrobial therapy
  * Treatment-limiting adverse event (AE) leading to discontinuation of study drug therapy, when subject required alternative antimicrobial therapy to treat the pneumonia
  * Death wherein pneumonia (ie,CABP) was considered causative
  Indeterminate: Inability to determine an outcome
Time Frame: 8 to 15 days after last dose of study drug
Population: The MITTE Population consisted of all subjects in the MITT Population (all randomized subjects who received any amount of the study drug) in PORT Risk Class III or IV. The Pneumonia Outcomes Research Team (PORT) scale of CAP severity in which Risk Class I is associated with the lowest risk for mortality and Risk Class V represents the highest risk.
Measure: Number; unit: participants
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Number analyzed (Participants) | 291 | 300
participants
  Clinical Cure | 244 | 233
  Clinical Failure | 34 | 58
  Indeterminate | 13 | 9
Statistical Analysis 1: Comparison: Ceftaroline Fosamil for Injection vs IV Ceftriaxone; The primary objective of this study was to determine the noninferiority in the clinical cure rate for ceftaroline compared to that for ceftriaxone at TOC in the CE and MITTE Populations in adult subjects with CABP; Test type: Non-Inferiority or Equivalence — A two-sided 95% Confidence Interval (CI) for the observed difference in the primary outcome measure (clinical cure rate) between the ceftaroline group and the ceftriaxone group was calculated based on each of the CE and the MITTE Populations at the TOC visit. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10% for each of the CE and MITTE Populations; Risk Difference (RD) = 6.2, 95% CI 2-sided [-0.2 to 12.6] — Risk difference corresponds to Ceftaroline clinical cure rate minus Ceftriaxone clinical cure rate. The confidence interval was calculated using the Miettinen and Nurminen method without adjustment

2. Secondary Outcome: Clinical Response at End of Therapy (EOT)
Time Frame: Last day of study drug administration
Reporting Status: Not Posted

3. Secondary Outcome: Microbiological Success Rate at Test of Cure (TOC)
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

4. Secondary Outcome: Overall (Clinical and Radiographic) Success Rate at Test of Cure (TOC)
Time Frame: 8-15 days after last day of study drug
Reporting Status: Not Posted

5. Secondary Outcome: Clinical and Microbiological Response by Pathogen at TOC
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Relapse at Late Follow Up (LFU)
Time Frame: 21-35 days after last dose of study drug
Reporting Status: Not Posted

7. Primary Outcome: Clinical Cure Rate for Ceftaroline Compared to That for Ceftriaxone at Test-of-Cure (TOC) in the Clinically Evaluable (CE) Population
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

8. Secondary Outcome: Microbiological Re-infection/Recurrence at LFU
Time Frame: 21 to 35 days after last dose of study drug
Reporting Status: Not Posted

9. Secondary Outcome: Evaluate Safety
Time Frame: first dose, throughout the treatment period, and up to the TOC visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety analysis was performed on the Safety Population, consisting of any subject who received any amount of actual study drug
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Serious Adverse Events (participants affected / at risk) | 28/298 | 33/308
Other Adverse Events (participants affected / at risk) | 65/298 | 53/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=298) | IV Ceftriaxone (N=308)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 2 (2) | 0 (0)
Multiorgan disorder (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 2 (2)
Pyothorax (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer, state unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=298) | IV Ceftriaxone (N=308)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 7 (7)
Headache (Nervous system disorders) | 10 (10) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 8 (8) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Phlebitis (Vascular disorders) | 7 (7) | 5 (5)
Hypertension (Vascular disorders) | 6 (6) | 8 (8)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No